CLINICAL TRIAL: NCT06893445
Title: The Effect of Deep Tissue Massage on Respiratory Parameters in People With Asthma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Bartosz Trybulec, Assistant professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 118.0043.1.81.2025
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Massage; Asthma Patients
Keywords: deep tissue massage; spirometry; asthma; respiratory parameters
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deep Tissue Massage Group (Experimental): The one session of deep tissue massage will be performed. The patient's positions will be changed depending on the specificity of used techniques. The following techniques will be used: • Shifting the rectus abdominis m., • Stretching of the fascia within the costal arches, • trigger points compression (30-60 s). • Stretching of the chest fascia, superficially with forearm or fingertips on intercostal muscles, • "filleting" the pectoral muscles, • "hook and stretch" with the proximal phalanges of the fingers 2-4 and the forearm • "filleting" between the pectoral muscles and the deltoids, • Releasing the lateral edge of the scapula using the fingers and stretching the tissues, Releasing the medial edge of the scapula using the fingers and the weight of the patient, • "hook and stretch" of the trapezius muscle, • Subsequently, the patient will take a prone position. • Stretching of the levator scapulae and supraspinatus muscles using the fist, forearm and elbow will be performed.
  Interventions: Procedure: Deep Tissue Massage
- Classic Massage Group (Active Comparator): The one session of classic massage will be performed. The massage will be performed with moderate force. The entire procedure will take about 15-20 min. The sequence of standard classic massage techniques will be used in standard way and patterns.
  Interventions: Procedure: Classic massage

INTERVENTIONS:
Procedure: Deep Tissue Massage — Administered as a soft tissue mobilization performed by the therapist with fingertips, knuckles, elbows and/or fists on the tissues that manifest symptoms of fascial restrictions. The techniques were performed with individually adjusted force until the change (eg. increased mobility) in the tissue being treated was stated by the therapist.
  Arms: Deep Tissue Massage Group
Procedure: Classic massage — The subject was lying supine on the table, with a roller placed under the knee joints, the upper limbs along the body. The following sequence of techniques was used in the longitudinal and transverse strands and in the intercostal spaces (excluding the breast in women): effleurage, friction, petrissage, pressures, tapotement and vibrations.
  Arms: Classic Massage Group

SUMMARY:
Bronchial asthma, as a chronic inflammatory disease of the respiratory tract, significantly reduces the quality of life of patients. Standard treatment includes pharmacotherapy, but a holistic approach, including manual therapies, can support pharmacological therapy, reducing the need for drugs.

The aim of the research is to verify whether deep tissue massage (DTM) techniques applied to the chest significantly affect respiratory parameters in people with asthma. The study is the next stage of the study conducted on healthy people. After obtaining positive results in the study involving people not suffering from respiratory diseases, the next step is to examine people with, in this case, bronchial asthma. It is important to determine whether the use of this form of manual therapy can bring benefits in the context of improving respiratory functions, reducing respiratory muscle tension and relieving subjective symptoms associated with asthma, such as shortness of breath or limitations in everyday functioning.

The hypothesis assumes that DTM techniques can have a bigger effect on the respiratory system than classic massage (CM).

The study is a randomized controlled trial, where participants will be randomly assigned to one of two groups: the study group (subjected to DTM) or the control group (subjected to CM). Before and after the massage intervention, participants will undergo spirometry to assess the changes in respiratory parameters. The obtained data will then be analyzed for effects on respiratory parameters and differences between both groups.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with bronchial asthma
* stable health condition, allowing participation in the study
* informed consent to participate in the study

Exclusion Criteria:

* acute or chronic comorbidities that may affect the results (e.g. COPD, heart failure, cancer)
* any chest surgery performed within the last 6 months
* contraindications to massage (e.g. skin infections, wounds)
* pregnancy
* participation in other clinical trials in the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of change of lung vital capacity | twice: before and immediately after procedure administration in both groups
  The vital capacity of the lungs will be assessed with spirometer. The subject stood with legs hip-width apart. For each measurement, disposable cardboard mouthpieces will be used. The examined person holds the device vertically with both hands. At the examiner's command, subject will take in as much air as possible, then tightly biet the mouthpiece with his mouth, and with all of their strength, exhale air into the device for as long as possible. The subject will have only 1 attempt-measured values were recorded with an accuracy of 50 mL.
Assessment of change of chest circumference | twice: before and immediately after procedure administration in both groups
  The chest circumference will be measured with a measuring tape, wrapped horizontally around the chest at the level of the xiphoid process. The subject stand with feet hip-width apart, arms hanging along the body. At the command, the subject will take a maximum breathe in (first measurement) and exhale to the maximum for the next (second measurement). Obtained values will be recorded with an accuracy of 0.5 cm.
Assessment of change of blood oxygen saturation | twice: before and immediately after procedure administration in both groups
  Testing blood oxygen saturation will be performed in a sitting position with digital pulseoximeter. The device will be put on the second finger of the left hand each time. The highest value displayed by the pulseoximeter within 30 s will be recorded with an accuracy of 1%.
Asessment of change of Peak Expiratory Flow (PEF) | twice: before and immediately after procedure administration in both groups
  Dynamic spirometry test will be performed with spirometer to assess the peak expiratory flow (PEF) measured in liters per second [l/s]. The subject will sit with his legs on the floor-hip joint flexed at an angle of 70o-90o and carry out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle will be performed at least 3 times obtaining 3 measurements and the mean value will be calculated.
Assessment of change of Forced Vital Capacity | twice: before and immediately after procedure administration in both groups
  The forced vital capacity (FVC), measured in liters will be assessed with spirometer. The subject will sit with his legs on the floor-hip joint flexed at an angle of 70o-90o and carry out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ".
Assessment of change of Maximum Expiratory Flow | twice: before and immediately after procedure administration in both groups
  Assessment of the maximum expiratory flow (MEF), measured in liters per second will be performed with spirometer. The subject will sit with his legs on the floor-hip joint flexed at an angle of 70o-90o and carry out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle will be performed at least 3 times obtaining 3 measurements and the mean value will be calculated.
Assessment of change of Forced Expiratory Volume in one second | twice: before and immediately after procedure administration in both groups
  Assessment of the forced expiratory volume in 1 s (FEV1) measured in literswill be performed with spirometer. The subject will sit with his legs on the floor-hip joint flexed at an angle of 70o-90o and carry out the following command: "Breathe calmly. On my command, breathe in as much as possible, as quickly as possible, as intensively as possible, and while at the top of the inhalation, without waiting, breathe out as hard and as long as possible ". This cycle will be performed at least 3 times obtaining 3 measurements and the mean value will be calculated.
Assessment of change of Maximum Voluntary Ventilation | twice: before and immediately after procedure administration in both groups
  Assessing the maximum voluntary ventilation (MVV) measured in liters per minute will be performed with spirometer. The subject will sit with his legs on the floor-hip joint flexed at an angle of 70o-90o and carried out the following command: "Breathe calmly. On my command, inhale and exhale as quickly and as deeply as possible for 15 s until you hear the 'stop' command. This cycle will be performed at least 3 times obtaining 3 measurements and the mean value will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz T Trybulec, PhD, Study Director — Jagiellonian University
Locations (2):
- Poland (2):
  - Department of Physiotherapy, Faculty of Health Sciences, Jagiellonian University Medical College, Krakow
  - The "Wieliczka" Salt Mine Health Resort, Wieliczka

IPD SHARING:
Plan to Share IPD: No
due to The General Data Protection Regulation directives